CLINICAL TRIAL: NCT02371343
Title: Effect of Fish Oil Supplementation in Women With Gestational Diabetes on Insulin Like Growth Factor-1 DNA Methylation in Newborns
Brief Title: Fish Oil Supplementation in Women With Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Dilek Dilli, Dilek Dilli, MD, Dr. Sami Ulus Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SamiUlusCH
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Fetal Macrosomia; Congenital Abnormality; Other Respiratory Problems After Birth
MeSH Terms: conditions — Fetal Macrosomia; Congenital Abnormalities | interventions — Fish Oils; Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish-Oil (Active Comparator): The pregnants with gestational diabetes given fish oil:
  (Ocean Plus, 1200 mg, EPA 384 mg DHA 252 mg, total omega-3 782 mg, 50 soft gel, Ocean®, German) During third trimester of pregnancy, Once in a day
  Interventions: Dietary Supplement: Fish oil, Ocean plus
- Sunflower oil (Placebo Comparator): The pregnants with gestational diabetes given sunflower oil:
  Sunflower oil capsules will be prepared in the pharmacy as the same size and colour with fish oil capsules During third trimester of pregnancy, Once in a day
  Interventions: Dietary Supplement: Sunflower Oil

INTERVENTIONS:
Dietary Supplement: Fish oil, Ocean plus — Ocean Plus, 1200 mg, EPA 384 mg DHA 252 mg, total omega-3 782 mg, 50 soft gel, Ocean®, Germany
  Arms: Fish-Oil
Dietary Supplement: Sunflower Oil
  Arms: Sunflower oil

SUMMARY:
Gestational diabetes is the development of diabetes during pregnancy. Left untreated, gestational diabetes and preeclampsia can lead to serious -- or even fatal -- complications for both mother and child. Some evidence suggesting omega-3 fatty acids might help protect women from two serious pregnancy complications -- gestational diabetes and preeclampsia. Omega-3 fatty acids, in particular Docosahexaenoic acid (DHA), help a pregnant woman give her developing baby every advantage in life starting in-utero. Recent studies suggested that the biologic processes underlying the observed associations may involve epigenetic changes, specifically DNA methylation. In this study the investigators aimed to examine the effect of fish oil supplementation in women with gestational diabetes mellitus on newborn outcomes and insulin like growth factor 1 DNA methylation.

DETAILED DESCRIPTION:
Gestational diabetes is the development of diabetes during pregnancy. According to the National Institutes of Health, gestational diabetes occurs in about 5 percent of all pregnancies in the United States, resulting in about 200,000 cases a year. Treatment involves dietary measures, exercise and, in some cases, insulin injections. All pregnant women should be taking a prescribed pre-natal vitamin, and should also supplement with fish oil or another source of omega-3 fatty acids to help support the nervous system of their developing child.

Left untreated, gestational diabetes and preeclampsia can lead to serious -- or even fatal -- complications for both mother and child. In diabetic pregnancies there is an increased risk of birth defects. Some evidence suggesting omega-3 fatty acids might help protect women from two serious pregnancy complications -- gestational diabetes and preeclampsia. Omega-3 fatty acids, in particular Docosahexaenoic acid (DHA), help a pregnant woman give her developing baby every advantage in life starting in-utero. In general the omega-3 fatty acids found in fish help the cardiovascular system, the brain (including moods), and even the brain and eyes of a developing baby. The risk of pre-term delivery and low birth weight is three and a half times higher when mothers are deficient in DHA. Recent studies suggested that the biologic processes underlying the observed associations may involve epigenetic changes, specifically DNA methylation. In this study the investigators aimed to examine the effect of fish oil supplementation in women with gestational diabetes mellitus on newborn outcomes and insulin like growth factor 1 DNA methylation.

ELIGIBILITY:
Inclusion Criteria:

* Women who were diagnosed as gestational diabetes mellitus (GDM) between 24 and 28th week of pregnancy
* Women with GDM and accepted to be participate in the study
* Women younger that 40 years old
* The newborns of the women with GDM

Exclusion Criteria:

* The history of Type 1 diabetes melitus
* Abnormal glucose tolerance <20th gestational week
* The history of chronic illness in the mother
* Women who eat fish <2 times in a week
* Any history of sea-food allergy in the mother

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Birth size | 1 year
  Birth size of the newborns

SECONDARY OUTCOMES:
Insulin like growth factor DNA methylation | 1 year
  Insulin like growth factor DNA methylation

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Dilli, Assoc Prof, Principal Investigator — Teaching assistant
Locations (1):
- Sami Ulus CH, Ankara, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Guermouche B, Soulimane-Mokhtari NA, Bouanane S, Merzouk H, Merzouk S, Narce M. Effect of dietary n - 3 polyunsaturated fatty acids on oxidant/antioxidant status in macrosomic offspring of diabetic rats. Biomed Res Int. 2014;2014:368107. doi: 10.1155/2014/368107. Epub 2014 Jun 2. PMID 24987679
- [Result] Soulimane-Mokhtari NA, Guermouche B, Yessoufou A, Saker M, Moutairou K, Hichami A, Merzouk H, Khan NA. Modulation of lipid metabolism by n-3 polyunsaturated fatty acids in gestational diabetic rats and their macrosomic offspring. Clin Sci (Lond). 2005 Sep;109(3):287-95. doi: 10.1042/CS20050028. PMID 15898958
- [Derived] Dilli D, Dogan NN, Ipek MS, Cavus Y, Ceylaner S, Dogan H, Dursun A, Kucukozkan T, Zenciroglu A. MaFOS-GDM trial: Maternal fish oil supplementation in women with gestational diabetes and cord blood DNA methylation at insulin like growth factor-1 (IGF-1) gene. Clin Nutr ESPEN. 2018 Feb;23:73-78. doi: 10.1016/j.clnesp.2017.12.006. Epub 2017 Dec 30. PMID 29460817